CLINICAL TRIAL: NCT03022136
Title: Observation Study of Thoracic Dermatomes
Brief Title: To Map Human Lower Thoracic Dermatomes by Epidural Block
Acronym: LTDEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Liu Yong, Principal Investigator, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Der-201701
Record Dates: First submitted 2017-01-10; First posted 2017-01-16 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Urological Disease; Anesthesia
Keywords: epidural block; dermatome; human; spinal nerve; thoracic
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epidural Block (Experimental): Epidural block for patients undergoing urological surgery
  Interventions: Other: cold sensation method

INTERVENTIONS:
Other: cold sensation method — Complete sensory loss to ice will be evaluated form anterior median line to posterior median line at the end of surgery.

SUMMARY:
Significant differences exist among various dermatome maps. In addition, there were no anatomical landmarks to evaluate the dermatome at the back. The investigators aim to map the sensory innervations of lower thoracic nerves and find the dorsal landmarks to evaluate sensory innervations by epidural block. Patients undergoing urological surgery will receive epidural block. Fifty patients with superior border of complete sensory loss to ice from T9 to T12 (anterior median line) will be included in this study. The sensory loss to ice will be evaluated at midclavicular line, anterior axillary line, posterior axillary line, scapular line and posterior median line. The level of vertebrae will be identified and marked by ultrasound. The superior border of complete sensory loss to ice from anterior median line to posterior median line will be recorded for every patient. The dermatome map of T9 to T12 will be drawn. The landmarks of sensory innervations at posterior median line will be established using vertebrae.

DETAILED DESCRIPTION:
Background: The tract for percutaneous nephrolithotomy is typically established in the 11th intercostal space or in the subcostal area. According to Keegan and Garrett's dermatome map, the somatic pain could be controlled if the 11th and 12th the spinal nerve been blocked. However, the investigators found that if the 11th and the 12th spinal nerve had been blocked by evaluating the landmarks of ventral landmarks (xiphoid process , umbilicus and pubic symphysis), the somatic pain of percutaneous nephrolithotomy could not be controlled. In order to find the reason, the investigators compared the four main dermatome maps created by Henry Head, Foerster, Keegan and Lee. There are significant differences of dermatome among these maps. In addition, there were no landmarks to evaluate the dermatome at the back.

Objectives: To map the sensory innervations of lower thoracic nerves and find the dorsal landmarks to evaluate sensory innervations by epidural block.

Methods: Adult patients undergoing elective percutaneous nephrolithotomy, ureteroscopic lithotripsy, transuretheral resection of prostate and transuretheral resection of bladder tumor will receive epidural block with 0.5% ropivacaine. Complete Sensory loss to ice will be evaluated at anterior median line as soon as the surgery was completed. The superior border of complete sensory loss to ice will be identified by ventral landmaks (xiphoid process , umbilicus and pubic symphysis). Fifty patients with superior border of complete sensory loss to ice from T9 to T12 will be included in this study. The sensory loss to ice will be evaluated at anterior median line, midclavicular line, anterior axillary line, posterior axillary line, scapular line and posterior median line. The level of vertebrae will be identified and marked by ultrasound. The superior border of complete sensory loss to ice form anterior median line to posterior median line will be drawn and recorded for every patient. The dermatome map from T9 to T12 will be drawn. The landmarks of sensory innervations at posterior median line will be established using vertebrae..

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for percutaneous nephtolithotomy, ureteroscopy lithotripsy, transurethral resection of bladder tumor or transurethral resection of the prostate
* American Society of Anesthesiologists physical statusⅠ-Ⅲ
* Informed consent

Exclusion Criteria:

* Coagulopathy, on anticoagulants
* History of surgery on spine
* Spine deformity
* A known allergy to the drugs being used
* Tumer or infection at the site of puncture
* refusal to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Superior border of sensory block was assessed by cold sensation method | at the end of surgery
  The sensory loss to ice will be evaluated at anterior median line, midclavicular line, anterior axillary line, posterior axillary line, scapular line and posterior median line. The level of vertebrae will be identified and marked by ultrasound. The upper border of complete sensory loss to ice form anterior median line to posterior median line will be drawn and recorded for every patient.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Liu, MD, Principal Investigator — Department of Anesthesiology,Tongji Hospital,Wuhan
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
Damatomes of sensory loss to cold of each patient. Investigators can contact us by e-mail.

REFERENCES:
- [Result] Head H, Campbell AW, Kennedy PG. The pathology of Herpes Zoster and its bearing on sensory localisation. Rev Med Virol. 1997 Sep;7(3):131-143. doi: 10.1002/(sici)1099-1654(199709)7:33.0.co;2-7. No abstract available. PMID 10398478
- [Result] Wolff AP, Wilder Smith OH, Crul BJ, van de Heijden MP, Groen GJ. Lumbar segmental nerve blocks with local anesthetics, pain relief, and motor function: a prospective double-blind study between lidocaine and ropivacaine. Anesth Analg. 2004 Aug;99(2):496-501, table of contents. doi: 10.1213/01.ANE.0000122268.70154.A9. PMID 15271730
- [Result] Greenberg SA. The history of dermatome mapping. Arch Neurol. 2003 Jan;60(1):126-31. doi: 10.1001/archneur.60.1.126. PMID 12533100
- [Result] Lee MW, McPhee RW, Stringer MD. An evidence-based approach to human dermatomes. Clin Anat. 2008 Jul;21(5):363-73. doi: 10.1002/ca.20636. PMID 18470936
- [Result] Downs MB, Laporte C. Conflicting dermatome maps: educational and clinical implications. J Orthop Sports Phys Ther. 2011 Jun;41(6):427-34. doi: 10.2519/jospt.2011.3506. Epub 2011 May 31. PMID 21628826
- [Result] Ladak A, Tubbs RS, Spinner RJ. Mapping sensory nerve communications between peripheral nerve territories. Clin Anat. 2014 Jul;27(5):681-90. doi: 10.1002/ca.22285. Epub 2013 Jul 3. PMID 23824984